CLINICAL TRIAL: NCT03552952
Title: Development of Preterm Infant Gut Microbiome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Other Study IDs: 0490-17-RMB CTIL
Record Dates: First submitted 2018-05-22; First posted 2018-06-12 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Premature Infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm infants: 100 preterm infants
  Interventions: Other: No intervention
- Term infants: 100 term healthy infants
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study aims to explore the developmental of the gut microbiome in preterm infants as they grow and mature

DETAILED DESCRIPTION:
Preterm birth, defined as childbirth occurring at less than 37 completed weeks, is a major determinant of neonatal mortality and morbidity and has long-term adverse consequences for health. The human microbiome is the collective genome of the immense ecosystem of trillions of microbes and is considered to have a coevolved relationship with the immune system and fundamental roles in multiple aspects of human physiology. Little is known about the developmental of the gut microbiome in preterm infants as they grow and mature.

One hundred premature infants born in Rambam healthcare campus in Haifa, Israel, will be recruited to the study and 100 term healthy infants will be recruited as controls. Infants born before 24 weeks of gestation or have birth weights of less than 400 g and infants with severe congenital anomalies will be excluded from the study. Fecal samples will be collected during the hospital stay and in follow-up visits. Blood samples will be taken during the hospital stay. The investigators will analyze the data from this clinical cohort using computational and experimental approaches for extracting novel information on microbiome composition and development, gene function, metabolic pathways and metabolite production.

ELIGIBILITY:
Inclusion Criteria:

* Premature and term infants born in Rambam healthcare campus in Haifa, Israel

Exclusion Criteria:

* Infants born before 24 weeks of gestation or have birth weights of less than 400 g and infants with severe congenital anomalies will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Premature and term infants
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-03-08 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbial abundance over time | One year
  Preterm infants and full-term infants fecal DNA at different time points

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neonatology and Neonatal Intensive Carer unit Rambam medical center, Haifa, Israel